CLINICAL TRIAL: NCT02459262
Title: A Two-part, Phase I, Randomised, Double-blind, Placebo-controlled, Parallel Group Study to Evaluate the Safety, Tolerability and Immunogenicity of a Dose Range og Group B Streptococcus Vaccine in Healthy Female Volunteers Aged 18 to 40.
Brief Title: Safety and Immunogenicity of a Group B Streptococcus Vaccine in Non-pregnant Women 18-40 Years of Age.
Acronym: MVX13211
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Minervax ApS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2014-004542-10
Record Dates: First submitted 2015-05-22; First posted 2015-06-02 (Estimated); Results first posted 2021-01-14 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2020-11

CONDITIONS: Infection by Streptococcus Group B

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GBS-NN Vaccine (Active Comparator): GBS-NN vaccine administered either adsorbed to Alhydrogel® or alone.
  Interventions: Biological: GBS-NN vaccine
- Sterile dilution buffer with Alhydrogel (Placebo Comparator): The placebo will contain either Alhydrogel® or buffer alone.
  Interventions: Biological: GBS-NN vaccine

INTERVENTIONS:
Biological: GBS-NN vaccine — Three dose levels will be administered, with and without Alhydrogel®

SUMMARY:
Part A: The primary objective is to evaluate the safety and tolerability of a potential vaccine against Group B streptococcus.

Part B: To evaluate the long term safety profile of the GBS-NN vaccine up to one year following the first dose.

DETAILED DESCRIPTION:
Part A: Subjects will receive 2 doses of the vaccine, GBS-NN, and will be followed for 12 weeks after the first dose of the vaccine. The following safety endpoints will be evaluated to support this objective: local and systemic reactogenicity; adverse events; laboratory tests; urinalysis; vital signs; 12-Lead ECG parameters; physical examination. In addition hereto, immunological parameters will be evaluated.

Part B: Subjects will receive one or 2 doses of GBS-NN, and will be followed for 12 months after the first dose of the vaccine. The following safety endpoints will be evaluated to support this objective: local and systemic reactogenicity; adverse events; laboratory tests; urinalysis; vital signs; 12-Lead ECG parameters; physical examination. In addition hereto, immunological parameters will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult female volunteers (as determined by medical history, physical examination, laboratory test values, vital signs and electrocardiograms [ECGs] at screening) aged 18 - 40 years.
2. Body mass index (BMI) ≥ 18 and ≤ 30 kg/m2.
3. Volunteers weight ≥ 50kg and ≤100kg at screening.
4. Able to voluntarily provide written informed consent to participate in the study.
5. Must understand the purposes and risks of the study and agree to follow the restrictions and schedule of procedures as defined in the protocol.
6. Volunteers must be pre-menopausal. Volunteers who have had a hysterectomy will have pre-menopausal status confirmed by a FSH and oestradiol test.
7. Females of childbearing potential must have a negative pregnancy test at screening (β HCG) and prior to each dose and must be willing to use an adequate and highly effective method of contraception until at least Day 85 of the study. A highly effective method of birth control is defined as one which results in a low failure rate (i.e. less than 1% per year) when used consistently and correctly such as sterilisation, implants, injectables, combined oral contraceptives, IUDs (Intrauterine Device), condoms, occlusive caps (cervical/vault caps) with spermicidal foam/gel/ film/cream/suppository. True sexual abstinence is acceptable when this is in line with the preferred and usual lifestyle of the volunteer (periodic abstinence e.g. calendar, ovulation, symptothermal, post-ovulation methods, declaration of abstinence for the duration of the trial, and withdrawal are not acceptable methods of contraception)
8. In Part A: Volunteers must be non-smokers for at least 3 months prior to first studyvaccine administration. In Part B: Volunteers may be light smokers i.e. up to a maximum of 5 cigarettes per day or nicotine equivalent.
9. Must be willing to consent to have data entered into The Over Volunteering Prevention System (TOPS).
10. The volunteer's primary care physician has confirmed within the last 12 months that there is nothing in their medical history that would preclude their enrolment into a clinical trial.

Exclusion Criteria:

1. Volunteers with history or presence of significant cardiovascular disease, pulmonary, hepatic, gallbladder or biliary tract, renal, haematological, gastrointestinal, endocrine, immunologic, dermatological, neurological, psychiatric, autoimmune disease or current infection.
2. Pregnant or lactating females.
3. Laboratory values at screening which are deemed to be clinically significant, unless agreed in advance by the Sponsor's Responsible Medic and Principal Investigator.
4. Current or history of drug or alcohol abuse, or a positive alcohol breath test prior to first dosing.
5. Positive for human immunodeficiency virus (HIV), hepatitis B or hepatitis C.
6. Participation in a clinical drug study during the 90 days preceding the initial dose in this study.
7. Any significant illness during the 4 weeks preceding check-in for this study (Day 1).
8. Volunteers with a history of severe allergic reactions after previous vaccination.
9. Volunteers who have received any vaccine within 30 days of screening, or who are planning to receive a vaccine up to Day 85 of the study.
10. Volunteers receiving immunosuppressive therapy (e.g. systemic steroids, cancer therapies, methotrexate, azathioprine) in the 6 months prior to screening, antibiotics within 10 days of receiving the first dose or taking any short-term medications including over-the-counter preparations, vitamins, herbal and/or mineral supplements within 7 days of the first dose. Chronic medications such as antihypertensives, bronchodilators, oral contraceptives or statins that do not affect the immune system, will be permitted and allowed to continue during the study at the discretion of the Investigator. Paracetamol will be permitted for the treatment of headache or other symptoms.
11. Volunteers with tattoos at the proposed site of vaccine administration.
12. Donation of blood or blood products within 90 days prior to vaccine administration.
13. Volunteers who, in the opinion of the Investigator, are unsuitable for participation in the study.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 240 (Actual)
Dates: Start 2015-05; Primary Completion 2017-04-12 (Actual); Study Completion 2017-04-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Per Fisher, PM/CEO, Study Director — MinervaX ApS, Ole Maaløes Vej 3, DK-2200 Copenhagen N, Denmark
Locations (1):
- Biokinetic Europ Ltd, Belfast, United Kingdom

REFERENCES:
- [Derived] Pawlowski A, Lannergard J, Gonzalez-Miro M, Cao D, Larsson S, Persson JJ, Kitson G, Darsley M, Rom AL, Hedegaard M, Fischer PB, Johansson-Lindbom B. A group B Streptococcus alpha-like protein subunit vaccine induces functionally active antibodies in humans targeting homotypic and heterotypic strains. Cell Rep Med. 2022 Feb 15;3(2):100511. doi: 10.1016/j.xcrm.2022.100511. eCollection 2022 Feb 15. PMID 35243418
- [Derived] Fischer P, Pawlowski A, Cao D, Bell D, Kitson G, Darsley M, Johansson-Lindbom B. Safety and immunogenicity of a prototype recombinant alpha-like protein subunit vaccine (GBS-NN) against Group B Streptococcus in a randomised placebo-controlled double-blind phase 1 trial in healthy adult women. Vaccine. 2021 Jul 22;39(32):4489-4499. doi: 10.1016/j.vaccine.2021.06.046. Epub 2021 Jun 30. PMID 34215454

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Part A: Healthy females were recruited to receive two doses of either GBS-NN vaccine with or without Alhydrogel® gel adjuvant at three dose levels (10mcg, 50mcg, 250mcg) or placebo.
  Part B: Doses of 50mcg (2 doses) and 100mcg (1 and 2 doses) were selected from the antibody levels at 8 weeks from Part A and vaccine was administered with Alhydrogel®. Participants were healthy females and did not include participants from Part A. They were followed up for 1 year.
Pre-assignment Details: Part A was the dose-finding part of the study and 60 healthy female participants received either 2 doses of GBS-NN 10mcg, 50mcg, 250mcg or placebo (4:1 ratio of active:placebo). Based on the 8 week (Day 57) antibody levels from Part A, 180 healthy female participants in Part B were recruited to receive either 2 doses of GBS-NN 50mcg, 2 doses of GBS-NN 100mcg, 1 dose of GBS-NN 100mcg or placebo (3:1 ratio of active to placebo). Participants in Part A were not allowed to participate In Part B.
Groups:
- Part A GBS-NN Vaccine 10mcg: GBS-NN 10mcg vaccine administered without Alhydrogel® by intramuscular injection on Day 1 and Day 29
- Part A GBS-NN Vaccine 50mcg: GBS-NN 50mcg vaccine administered without Alhydrogel® by intramuscular injection on Day 1 and Day 29
- Part A GBS-NN Vaccine 250mcg: GBS-NN 250mcg vaccine administered without Alhydrogel® by intramuscular injection on Day 1 and Day 29
- Part A GBS-NN 10mcg Vaccine Administered With Alhydrogel® Adjuvant: GBS-NN 10mcg vaccine administered with Alhydrogel® by intramuscular injection on Day 1 and Day 29
- Part A GBS-NN 50mcg Vaccine Administered With Alhydrogel® Adjuvant; Part B GBS-NN Vaccine 50mcg: GBS-NN 50mcg vaccine administered with Alhydrogel® by intramuscular injection on Day 1 and Day 29
- Part A GBS-NN 250mcg Vaccine Administered With Alhydrogel® Adjuvant: GBS-NN 250mcg vaccine administered with Alhydrogel® by intramuscular injection on Day 1 and Day 29
- Part A Placebo: Alhydrogel® mixed with dilution buffer or buffer alone administered by intramuscular injection
- Part B GBS-NN Vaccine 100mcg 2 Dose Regimen: GBS-NN 100mcg vaccine administered with Alhydrogel® by intramuscular injection on Day 1 and Day 29
- Part B GBS-NN Vaccine 100mcg Single Dose: GBS-NN 100mcg vaccine administered with Alhydrogel® by intramuscular injection on Day 1
- Part B Placebo: Alhydrogel® mixed with dilution buffer and administered by intramuscular injection
Period: Overall Study
Arm/Group | Part A GBS-NN Vaccine 10mcg | Part A GBS-NN Vaccine 50mcg | Part A GBS-NN Vaccine 250mcg | Part A GBS-NN 10mcg Vaccine Administered With Alhydrogel® Adjuvant | Part A GBS-NN 50mcg Vaccine Administered With Alhydrogel® Adjuvant | Part A GBS-NN 250mcg Vaccine Administered With Alhydrogel® Adjuvant | Part A Placebo | Part B GBS-NN Vaccine 50mcg | Part B GBS-NN Vaccine 100mcg 2 Dose Regimen | Part B GBS-NN Vaccine 100mcg Single Dose | Part B Placebo
Started | 8 | 8 | 8 | 8 | 8 | 8 | 12 | 45 | 45 | 45 | 45
Completed | 8 | 8 | 8 | 8 | 8 | 8 | 12 | 45 | 45 | 44 | 45
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part A GBS-NN Vaccine 10mcg With Alhydrogel® Adjuvant: GBS-NN 10 mcg vaccine administered with Alhydrogel® by intramuscular injection on Day 1 and Day 29
- Part A GBS-NN Vaccine 50mcg With Alhydrogel® Adjuvant; Part B GBS-NN Vaccine 50mcg: GBS-NN 50mcg vaccine administered with Alhydrogel® by intramuscular injection on Day 1 and Day 29
- Part A GBS-NN Vaccine 250mcg With Alhydrogel® Adjuvant: GBS-NN 250mcg vaccine administered with Alhydrogel® by intramuscular injection on Day 1 and Day 29
- Part B GBS-NN Vacine 100mcg 2 Dose Regimen: GBS-NN 100mcg vaccine administered with Alhydrogel® by intramuscular injection on Day 1 and Day 29
- Part B GBS-NN Vacine 100mcg Single Dose: GBS-NN 100mcg vaccine administered with Alhydrogel® by intramuscular injection on Day 1
- Total: Total of all reporting groups
Arm/Group | Part A GBS-NN Vaccine 10mcg | Part A GBS-NN Vaccine 50mcg | Part A GBS-NN Vaccine 250mcg | Part A GBS-NN Vaccine 10mcg With Alhydrogel® Adjuvant | Part A GBS-NN Vaccine 50mcg With Alhydrogel® Adjuvant | Part A GBS-NN Vaccine 250mcg With Alhydrogel® Adjuvant | Part A Placebo | Part B GBS-NN Vaccine 50mcg | Part B GBS-NN Vacine 100mcg 2 Dose Regimen | Part B GBS-NN Vacine 100mcg Single Dose | Part B Placebo | Total
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 12 | 45 | 45 | 45 | 45 | 240
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.6 (4.8) | 29.3 (6.6) | 30.4 (5.0) | 28.3 (7.4) | 31.3 (4.5) | 30.4 (5.7) | 28.5 (6.6) | 29.0 (6.3) | 30.3 (6.0) | 29.4 (6.5) | 28.7 (6.5) | 29.5 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 8 | 8 | 8 | 8 | 12 | 45 | 45 | 45 | 45 | 240
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 8 | 8 | 8 | 8 | 8 | 8 | 12 | 45 | 45 | 45 | 44 | 239
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 8 | 8 | 8 | 8 | 8 | 8 | 12 | 45 | 45 | 45 | 44 | 239
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 8 | 8 | 8 | 8 | 8 | 8 | 12 | 45 | 45 | 45 | 45 | 240

OUTCOME MEASURES:

1. Primary Outcome: Part A Number of Participants With Treatment Emergent Adverse Events
Description: Number of Participants with Treatment Emergent Adverse Events
Time Frame: 12 weeks (to Day 85)
Measure: Number; unit: participants
Arm/Group | Part A GBS-NN Vaccine 10mcg | Part A GBS-NN Vaccine 50mcg | Part A GBS-NN Vaccine 250mcg | Part A GBS-NN Vaccine 10mcg With Alhydrogel® Adjuvant | Part A GBS-NN Vaccine 50mcg With Alhydrogel® Adjuvant | Part A GBS-NN Vaccine 250mcg With Alhydrogel® Adjuvant | Part A Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 12
participants | 6 | 5 | 5 | 6 | 8 | 8 | 11

2. Primary Outcome: Part B Number of Participants With Treatment Emergent Adverse Events
Description: Number of Participants with Treatment Emergent Adverse Events
Time Frame: 12 weeks (to Day 85)
Measure: Number; unit: participants
Arm/Group | Part B GBS-NN Vaccine 50mcg | Part B GBS-NN Vacine 100mcg 2 Dose Regimen | Part B GBS-NN Vacine 100mcg Single Dose | Part B Placebo
Number analyzed (Participants) | 45 | 45 | 45 | 45
participants | 41 | 39 | 31 | 37

3. Secondary Outcome: Part A Antibody Concentration
Description: Geometric mean antibody concentration
Time Frame: 12 weeks (Day 85)
Measure: Geometric Mean (Full Range); unit: mcg/mL
Arm/Group | Part A GBS-NN Vaccine 10mcg | Part A GBS-NN Vaccine 50mcg | Part A GBS-NN Vaccine 250mcg | Part A GBS-NN Vaccine 10mcg With Alhydrogel® Adjuvant | Part A GBS-NN Vaccine 50mcg With Alhydrogel® Adjuvant | Part A GBS-NN Vaccine 250mcg With Alhydrogel® Adjuvant | Part A Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 12
mcg/mL | 1.977 [0.021 to 35.80] | 2.926 [0.27 to 17.40] | 7.195 [0.865 to 106] | 16.864 [1.11 to 263] | 14.999 [2.95 to 83.00] | 25.431 [0.59 to 277] | 0.199 [0.03 to 1.61]
Statistical Analysis 1: Comparison: Part A GBS-NN Vaccine 10mcg vs Part A GBS-NN Vaccine 50mcg vs Part A GBS-NN Vaccine 250mcg vs Part A GBS-NN Vaccine 10mcg With Alhydrogel® Adjuvant vs Part A GBS-NN Vaccine 50mcg With Alhydrogel® Adjuvant vs Part A GBS-NN Vaccine 250mcg With Alhydrogel® Adjuvant vs Part A Placebo; The objectives for Part A were to evaluate the effect of adjuvant and to inform the selection of dose levels for Part B. The study was not powered for inter-group comparisons; Test type: Other — ANOVA repeated measures: In-transformed antibody concentrations as dependent variable; dose level, time, presence of adjuvant and dose*time interaction as fixed effects; subjects as random effects; p = 0.0193, ANOVA — Adjuvant effect at Day 85, the primary immunological endpoint; Adjuvant effect, with higher antibody concentration values after all dose levels of vaccine was significant at all time points (D29, D43, D57, Day 85)

4. Secondary Outcome: Part B Antibody Concentration
Description: Geometric mean antibody concentration
Time Frame: 12 weeks (Day 85)
Measure: Geometric Mean (Full Range); unit: mcg/mL
Arm/Group | Part B GBS-NN Vaccine 50mcg | Part B GBS-NN Vacine 100mcg 2 Dose Regimen | Part B GBS-NN Vacine 100mcg Single Dose | Part B Placebo
Number analyzed (Participants) | 45 | 45 | 43 | 45
mcg/mL | 16.914 [0.90 to 247.00] | 15.459 [0.35 to 314.00] | 3.035 [0.17 to 50.20] | 0.234 [0.03 to 15.80]
Statistical Analysis 1: Comparison: Part B GBS-NN Vaccine 50mcg vs Part B GBS-NN Vacine 100mcg 2 Dose Regimen vs Part B GBS-NN Vacine 100mcg Single Dose vs Part B Placebo; Test type: Other; p < 0.0001, ANOVA

5. Secondary Outcome: Part B Antibody Concentration
Description: Geometric mean antibody concentration
Time Frame: 1 year (Day 365)
Measure: Geometric Mean (Full Range); unit: mcg/mL
Arm/Group | Part B GBS-NN Vaccine 50mcg | Part B GBS-NN Vacine 100mcg 2 Dose Regimen | Part B GBS-NN Vacine 100mcg Single Dose | Part B Placebo
Number analyzed (Participants) | 45 | 45 | 43 | 45
mcg/mL | 4.201 [0.24 to 58.40] | 5.934 [0.20 to 314.00] | 1.596 [0.06 to 117.00] | 0.263 [0.03 to 50.50]
Statistical Analysis 1: Comparison: Part B GBS-NN Vaccine 50mcg vs Part B GBS-NN Vacine 100mcg 2 Dose Regimen vs Part B GBS-NN Vacine 100mcg Single Dose vs Part B Placebo; Test type: Other; p < 0.0001, ANOVA

6. Secondary Outcome: Part B Number of Participants With Treatment Emergent Adverse Events
Description: Number of Participants with Treatment Emergent Adverse Events
Time Frame: Day 85 to Day 365
Measure: Number; unit: participants
Arm/Group | Part B GBS-NN Vaccine 50mcg | Part B GBS-NN Vacine 100mcg 2 Dose Regimen | Part B GBS-NN Vacine 100mcg Single Dose | Part B Placebo
Number analyzed (Participants) | 45 | 45 | 45 | 45
participants | 16 | 23 | 22 | 21

ADVERSE EVENTS:
Time Frame: Part A: to 12 weeks (D85) Part B: to 12 weeks (D85)
Arm/Group | Part A GBS-NN Vaccine 10mcg | Part A GBS-NN Vaccine 50mcg | Part A GBS-NN Vaccine 250mcg | Part A GBS-NN Vaccine 10mcg With Alhydrogel® Adjuvant | Part A GBS-NN Vaccine 50mcg With Alhydrogel® Adjuvant | Part A GBS-NN Vaccine 250mcg With Alhydrogel® Adjuvant | Part A Placebo | Part B GBS-NN Vaccine 50mcg | Part B GBS-NN Vacine 100mcg 2 Dose Regimen | Part B GBS-NN Vacine 100mcg Single Dose | Part B Placebo
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/12 | 0/45 | 0/45 | 0/45 | 0/45
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/12 | 0/45 | 0/45 | 0/45 | 1/45
Other Adverse Events (participants affected / at risk) | 6/8 | 5/8 | 5/8 | 6/8 | 8/8 | 8/8 | 11/12 | 41/45 | 39/45 | 31/45 | 37/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A GBS-NN Vaccine 10mcg (N=8) | Part A GBS-NN Vaccine 50mcg (N=8) | Part A GBS-NN Vaccine 250mcg (N=8) | Part A GBS-NN Vaccine 10mcg With Alhydrogel® Adjuvant (N=8) | Part A GBS-NN Vaccine 50mcg With Alhydrogel® Adjuvant (N=8) | Part A GBS-NN Vaccine 250mcg With Alhydrogel® Adjuvant (N=8) | Part A Placebo (N=12) | Part B GBS-NN Vaccine 50mcg (N=45) | Part B GBS-NN Vacine 100mcg 2 Dose Regimen (N=45) | Part B GBS-NN Vacine 100mcg Single Dose (N=45) | Part B Placebo (N=45)
Spontaneous abortion (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A GBS-NN Vaccine 10mcg (N=8) | Part A GBS-NN Vaccine 50mcg (N=8) | Part A GBS-NN Vaccine 250mcg (N=8) | Part A GBS-NN Vaccine 10mcg With Alhydrogel® Adjuvant (N=8) | Part A GBS-NN Vaccine 50mcg With Alhydrogel® Adjuvant (N=8) | Part A GBS-NN Vaccine 250mcg With Alhydrogel® Adjuvant (N=8) | Part A Placebo (N=12) | Part B GBS-NN Vaccine 50mcg (N=45) | Part B GBS-NN Vacine 100mcg 2 Dose Regimen (N=45) | Part B GBS-NN Vacine 100mcg Single Dose (N=45) | Part B Placebo (N=45)
Injection site pain (General disorders) | 1 | 1 | 1 | 6 | 4 | 4 | 4 | 26 | 26 | 16 | 18
Headache (Nervous system disorders) | 0 | 3 | 1 | 2 | 2 | 1 | 4 | 14 | 9 | 6 | 11
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 3 | 2 | 3 | 2 | 1
Nasopharyngitis (Infections and infestations) | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 15 | 7 | 12 | 5
Dysmenorrhoea (Reproductive system and breast disorders) | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 2 | 1 | 2
Seasonal allergy (Immune system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 2 | 2 | 1 | 4
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Injection site reaction (General disorders) | 0 | 0 | 1 | 2 | 6 | 2 | 2 | 2 | 2 | 0 | 5
Injection site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 2 | 2 | 3
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 3
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 2 | 2 | 0
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 3 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-11-30): https://cdn.clinicaltrials.gov/large-docs/62/NCT02459262/Prot_SAP_000.pdf